CLINICAL TRIAL: NCT01789918
Title: TrAnsCatHeter Intravascular Ultrasound Energy deliVery for rEnal Denervation
Brief Title: TrAnsCatHeter Intravascular Ultrasound Energy deliVery for rEnal Denervation (ACHIEVE)
Acronym: ACHIEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0030-HT
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Resistant Hypertension
Keywords: Hypertension; Blood pressure; Renal denervation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Percutaneous renal denervation (Experimental): PARADISE percutaneous renal denervation
  Interventions: Device: PARADISE percutaneous renal denervation

INTERVENTIONS:
Device: PARADISE percutaneous renal denervation — Intravascular ultrasound emission
  Other Names: ReCor Medical PARADISE

SUMMARY:
The ACHIEVE study is a single-arm, open-label, prospective, post-market follow-up study to include up to one hundred (100) eligible patients as defined within the clinical investigational plan, with a twelve month follow-up period. The ACHIEVE study was originally designed in accordance with the 2007 ESH ESC guidelines for resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Resistant hypertension, as defined in the 2007 ESH-ESC guidelines
* 18 years of age or older
* Negative pregnancy test for female patients of childbearing potential
* Willing and able to comply with follow-up requirements
* Signed informed consent

Exclusion Criteria:

* Secondary hypertension
* Main renal arteries length < 20 mm
* Main renal arteries diameter < 4 mm
* Renal artery stenosis
* Iliac/femoral artery stenosis precluding insertion of the catheter
* Untreated allergy to contrast media
* Currently participating in the study of an investigational drug or device
* Moderate to severe renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-01-09 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with device- or procedure-related adverse events | 12 months
  Anticipated adverse events include:
  * Access site and access-related vascular injury
  * Renal artery complications, including: stenosis, aneurysm, dissection, and perforation
  * Renal complications, including: renal infarction, acute kidney injury, and renal failure
  * Arterial and venous thromboembolic events, including: myocardial infarction, stroke or transient ischemic attack, pulmonary embolism, and deep vein thrombosis
  * Systemic effects, including: allergic reaction and infection
Change from baseline in systolic blood pressure | 12 months
  Change from baseline in systolic blood pressure

SECONDARY OUTCOMES:
Change from baseline in diastolic blood pressure | 12 months
  Change from baseline in diastolic blood pressure
Change from baseline in anti-hypertensive medication intake | 12 months
  Change from baseline in anti-hypertensive medication intake
Changes from baseline in pulse pressure and nocturnal dipping | 12 months
  Changes from baseline in pulse pressure and nocturnal dipping

OTHER OUTCOMES:
Change from baseline in EQ-5D Quality of Life score | 12 months
  Change from baseline in EQ-5D Quality of Life score
Change from baseline in cardiac function | 12 months
  Change from baseline in cardiac function

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, Professor, Principal Investigator — Universitäts-Herzzentrum Freiburg • Bad Krozingen
Locations (8):
- Germany (6):
  - Universitäts-Herzzentrum Freiburg • Bad Krozingen, Bad Krozingen
  - Universitätsklinikum Essen, Essen
  - CardioVasculäres Centrum, Frankfurt
  - Asklepios Klinik St. Georg, Hamburg
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Universitätsklinikum Lübeck, Lübeck
- Erasmus MC - Thoraxcenter, Rotterdam, Netherlands
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden